CLINICAL TRIAL: NCT05253079
Title: Erector Spinae Plane Block Versus Subcostal Transversus Abdominis Plane Block in Patients Undergoing Open Liver Resection Surgery: A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Subcostal Transversus Abdominis Plane Block in Open Liver Resection Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS-481-2021
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Analgesia; Hepatic Resection Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subcostal transversus abdominis plane block group (Active Comparator): subcostal transversus abdominis plane block
  Interventions: Other: subcostal transversus plane block
- erector spinae plane block group (Active Comparator): erector spinae plane block
  Interventions: Other: erector spinae plane block

INTERVENTIONS:
Other: subcostal transversus plane block — Patient in TAP block group will receive oblique subcostal TAP while in supine position using a linear 6-13 MHz ultrasound transducer. The operator will place the ultrasound probe obliquely on the upper abdominal wall along the subcostal margin near the xiphisternum of the sternum in the midline of the abdomen. The landmarks, which included the rectus abdominis muscle and underlying transversus abdominis muscle, will be identified near the costal margin and xyphoid. The probe will be then moved laterally until the aponeurosis of the external, internal oblique, and transversus abdominis are seen, and then the probe will be moved further laterally until the transversus abdominis muscle is identified. The operator will direct the needle toward the transversus abdominis, and the local anesthetic solution will be injected after negative aspiration between the rectus abdominis and transversus abdominis muscles along the subcostal line (in-plane superomedial to inferolateral)
  Arms: subcostal transversus abdominis plane block group
Other: erector spinae plane block — Patients in ESPB group will be turned to the lateral position and receive ESPB at the level of the 7th thoracic (T7) transverse process using a linear 6-13 MHz ultrasound transducer. The transducer will be positioned vertically 3 cm to the side of the midline to visualize the muscles of the back, the transverse process, and the pleura between the two transverse processes. Then, a 22G 10-mm needle will be introduced in the cranial-caudal direction toward the transverse process (T7) using the in-plane method till the needle tip crosses all the muscles. The tip of needle should be in the plane between the transverse process and the erector spinae muscle. After ensuring negative aspiration, the local anesthetic solution will be injected below the muscle. the procedure will be repeated on the other side
  Arms: erector spinae plane block group

SUMMARY:
Liver resection surgery is a common surgical procedure which is performed on patients with benign, malignant or metastatic hepatic tumor as well as for living liver donor. Liver resection surgery is usually performed through either right subcostal or inversed L-shaped incision; both approaches are associated with a significant postoperative pain which requires intensive analgesic plan to facilitate early mobilization and minimize complications.

There are various lines for pain management in liver resection surgery such as systemic analgesic drugs, neuraxial blocks (e.g., thoracic epidural analgesia) and transversus abdominis plane [TAP] block).

Systemic analgesic drugs are nearly constantly used in liver resection. However, being systemically administered, these drugs have many side effects on many organs and cannot totally eliminate postoperative pain. Thoracic epidural block is commonly associated with hypotension; furthermore, its use has other limitations such as delaying postoperative mobilization and possible hematoma and cord compression in patients with coagulopathy which is expected following liver resection. Therefore, there had been an increased interest in the use of abdominal field blocks to avoid disadvantages of neuraxial blocks and minimize the use of parenteral analgesic drugs.

TAP block is one of the classic field blocks which is extensively used in laparotomies including liver resection. However, the lack of visceral pain control TAP block influences the quality of its analgesic effect in this type of patients. Nevertheless, TAP block, namely the subcostal approach, is still the recommended field block in the latest procedure-specific recommendations for pain management in liver resection as it is the only block which showed good evidence.

In recent years, there has been increased interest in a newer field block, the erector spinae plane block (ESPB), due its easy performance and the possible coverage of visceral pain in addition to the somatic pain. ESPB showed promising results in liver resection surgery. ESBP was superior to TAP block in various abdominal surgeries. However, its analgesic efficacy had not been previously compared in relation to TAP in patients undergoing open liver resection surgery.

DETAILED DESCRIPTION:
An independent research assistant will be responsible for opening the envelope and drug preparation with no further involvement in the study. The local anesthetic solution preparation will be as follow; 2 syringes of 20 ml of 0.25% isobaric bupivacaine.

Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and pre-medication drugs will be delivered (metoclopramide 10 mg, and omeprazole 40 mg).

General anesthesia will be induced by 2-3 mg/kg propofol and 1-2 mcg/kg fentanyl. Tracheal intubation by direct laryngoscopy will be facilitated by atracurium 0.5 mg/kg. Anesthesia will be maintained by 2-2.5% sevoflurane and 0.1 mg/kg/20min atracurium.

After induction of anesthesia, patients will receive their assigned intervention.

Intraoperative analgesic management Morphine boluses (titrated 0.05 mg/kg boluses till response) will be given in case of inadequate analgesia (heart rate/mean blood pressure increase by 20% from the baseline) Intraoperative fluid and hemodynamic management will be according to the discretion of the attending anesthetist.

At the end of the surgery, all patients will receive intravenous paracetamol (1 g) and ketorolac (30 mg) before the extubation.

Postoperative care All patients will receive regular intravenous paracetamol 1 g/6hours and ketorolac 30 mg/8hours. Pain assessments using Numerical Rating Scale (NRS) will be performed at rest and during cough at 0.5, 1, 2, 4, 6, 18, 24 hours after leaving the operating room. If NRS score is > 3 intravenous titration of 2 mg morphine is given slowly to be repeated after 30 minutes if pain persisted. If other opioids are given, morphine equivalent dose will be calculated using opioids conversion chart.

Intravenous ondansetron 4 mg will be given to treat nausea or vomiting if occurs.

the following data will be recorded Complications: hematoma, nausea, vomiting, itching, urine retention, constipation, Initial pathology, type and length of skin incision, duration of surgery, blood loss, need for blood transfusion, vasoactive drugs Age, sex, American society of anesthesiologist-physical status (ASA), comorbidity, weight, height and body mass index

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years),
* ASA-physical status I-III
* undergoing open liver resection surgery for either primary/metastatic hepatic malignancy, biliary tract malignancy, or benign hepatic tumor

Exclusion Criteria:

* history of allergy to any of the study drugs,
* a body mass index (BMI) <18 or ≥ 35 kg/m2,
* coagulopathy (INR >1.5 and/or platelet count <70000/µL),
* local infection,
* history of chronic pain or regular opioid use;
* inability to comprehend the Numeric Rating Scale (NRS),
* liver resection combined with a second surgical procedure, laparoscopic resections,
* pregnant or lactating women.
* Patients with complicated procedures
* those needing postoperative ventilation will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
total morphine requirement in the first 24 hours | 0.5 hour after extubation till 24 hour after extubation
  mg

SECONDARY OUTCOMES:
intraoperative morphine requirement | 15 minutes after block administration till 1 minutes after extubation
  mg
time to first morphine requirement | 1 minute after block administration till 24 hours postoperatively
  hours
NRS | 0.5, 1, 2, 4, 6, 18, 24 hours after leaving the operating room
  11-points scale in which the patients are asked to circle the number between 0 and 10 that best describe their pain intensity. Zero represents 'no pain at all' whereas 10 represents 'the worst pain ever possible
Time to independent movement | 0.5 hour after extubation till 24 hour after extubation
  time in hours of being able to be independently mobile e.g. using the bathroom
heart rate | 15 minutes before induction of anesthesia, 15 minutes after induction of anesthesia, every 15 minutes intraoperatively and 0.5, 1, 2, 4, 6, 18, 24 hours postoperatively
  beat per minutes
mean arterial pressure | 15 minutes before induction of anesthesia, 15 minutes after induction of anesthesia, every 15 minutes intraoperatively and 0.5, 1, 2, 4, 6, 18, 24 hours postoperatively
  mmHg
Modified Ramsay Sedation Score | 0.5, 1, 2, 4, 6, 18, 24 hours after leaving the operating room
  1 = Awake and alert 2 = Slightly sedated, 3 = moderately sedated follows simple commands, 4 = deeply sedated, responds to nonpainful stimuli, 5 = deeply sedated, responds to painful stimuli, 6 = deeply sedated, unresponsive to painful stimuli

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data can be available from the principle investigator upon reasonable request

REFERENCES:
- [Derived] Mostafa M, Mousa MS, Hasanin A, Arafa AS, Raafat H, Ragab AS. Erector spinae plane block versus subcostal transversus abdominis plane block in patients undergoing open liver resection surgery: A randomized controlled trial. Anaesth Crit Care Pain Med. 2023 Feb;42(1):101161. doi: 10.1016/j.accpm.2022.101161. Epub 2022 Sep 22. PMID 36154912